CLINICAL TRIAL: NCT04243135
Title: Effects of Radial Extracorporeal Shock Wave Therapy (r-ESWT) on Clinical Variables and Isokinetic Performance in Patients With Knee Osteoarthritis
Brief Title: r-ESWT in Moderate Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Mustafa Turgut Yildizgoren, Principal Investigator, Clinical Assoc. Professor, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol Code: 2017/166
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Orthopedic Disorder
Keywords: r-ESWT; knee osteoarthritis; pain; function
MeSH Terms: conditions — Musculoskeletal Diseases; Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESWT group (Active Comparator): All patients in both groups were applied with a hot pack for 40-minutes, transcutaneous electrical nerve stimulation for 30-minutes (100 Hz frequency and 60 milliseconds pulse duration), and a home-based exercise program around the knee for 30-minutes per day for three weeks. Also, each patient in group 1 received shockwaves of continuous frequency and intensity (2000 shocks, 10 Hz, 2.0 to 3.0 bar), while the second group of patients received sham-ESWT. In group 1, for a total of 3 weeks, r-ESWT was undertaken with 2000 pulse each time at a week interval totaling 6000 pulse by using a radial shock wave therapy system (vibrolith ortho tip ESWT (ELMED Turkey)).
  Interventions: Device: ESWT
- Sham-ESWT group (Sham Comparator): The other group received sham-ESWT at 0.1 bar in the same area. The patients were placed supine with the affected knee at 90 degrees flexion at each treatment session. The shock wave probe was held stationary on painful points around the knee or at the patellofemoral and tibiofemoral borders of the target knee.
  Interventions: Device: ESWT

INTERVENTIONS:
Device: ESWT — Extracorporeal shock wave therapy

SUMMARY:
This study aims to compare the efficacy of r-ESWT treatment with sham-ESWT on pain, walking speed, physical function, and isokinetic muscle strength in knee osteoarthritis.

DETAILED DESCRIPTION:
Extracorporeal shock wave therapy (ESWT) has been increasingly used to help relieve pain and to remedy musculoskeletal disorders in recent years. ESWT seems to be an effective treatment modality many different musculoskeletal conditions, including rotator cuff tendinopathies, calcifying tendinopathy of the shoulder, lateral epicondylitis, greater trochanteric pain syndrome, patellar tendinopathy, achilles tendinopathy, plantar fasciitis, and bone disorders. ESWT seems to have chondroprotective, anti-inflammatory, neovascularization, anti-apoptotic, and tissue regeneration effect on tissues which could be relevant in the treatment of OA.

ELIGIBILITY:
Inclusion Criteria:

* Knee OA according to American College of Rheumatology (ACR) diagnostic criteria with Kellgren - Lawrence (K-L) grade 2 or 3.

Exclusion Criteria:

* Patients with secondary OA,
* severe chronic illness,
* poor general health status (heart failure, chronic bronchitis, etc.),
* chronic inflammatory diseases,
* knee replacement surgery,
* prior malignancy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | up to 12 weeks
  The VAS is used to measure and monitor pain intensity. Scores range from the absence of pain (0) to intolerable pain (0 or 10)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | up to 12 weeks
  Pain, joint stiffness, and physical functions were evaluated by the Western Ontario and McMaster Osteoarthritis Index (WOMAC). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
20-meter walk test | up to 12 weeks
  change from baseline on walking speed
isokinetic muscle performance | up to 12 weeks
  Isokinetic muscle performance was measured using a calibrated isokinetic test device named Humac®/NormTM Testing & Rehabilitation System (Computer Sports Medicine Inc. Stoughton, MA, USA). The knee extensor/flexor muscle group isokinetic muscle strength [peak torque (PT)] of both groups was evaluated using a calibrated isokinetic dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Uysal, MD, Principal Investigator — Mustafa Kemal University Medical School
Locations (1):
- Mustafa Kemal University, Hatay, Turkey (Türkiye)

REFERENCES:
- [Derived] Uysal A, Yildizgoren MT, Guler H, Turhanoglu AD. Effects of radial extracorporeal shock wave therapy on clinical variables and isokinetic performance in patients with knee osteoarthritis: a prospective, randomized, single-blind and controlled trial. Int Orthop. 2020 Jul;44(7):1311-1319. doi: 10.1007/s00264-020-04541-w. Epub 2020 Mar 26. PMID 32215674